CLINICAL TRIAL: NCT00074490
Title: Allogeneic HSCT Without Preparative Chemotherapy or With Low-Intensity Preparative Chemotherapy Using Sirolimus and Sirolimus-Generated Donor Th2 Cells for Therapy of Refractory Leukemia, Lymphoma, Myeloma, or Myelodysplastic Syndrome
Brief Title: Donor Stem Cell Transplant With No or Low-Intensity Chemotherapy Using Sirolimus and Treated Immune Cells to Treat Blood and Lymph Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Premature closure due to inability to accrue to ARM IVD, cohorts 1 and 2
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Pavletic, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040055; 04-C-0055; NCT00077480 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2003-12-15 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Lymphoma; Leukemia; Myeloproliferative Disorders; Multiple Myleoma; Myelodysplastic Syndrome
Keywords: Leukemia; Lymphoma; Multiple Myeloma; Bone Marrow Transplantation; Immune Therapy
MeSH Terms: conditions — Lymphoma; Leukemia; Myeloproliferative Disorders; Myelodysplastic Syndromes; Multiple Myeloma | interventions — Rituximab; fludarabine; fludarabine phosphate; Etoposide; Doxorubicin; liposomal doxorubicin; Vincristine; Cyclophosphamide; Transplantation; Prednisone; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm IVD cohort 1 (Th2 DLI) (Experimental): Patients receive low intensity fludarabine phosphate intravenous (IV) and cyclophosphamide IV on days -6 to -3. Patients undergo donor lymphocyte infusion (DLI) with sirolimus generated donor T-helper 2 (Th2) cells on day 14 (single T-Rapa cell DLI in patients with cluster of differentiation 4 (CD4) count between 100 and 200 inclusive)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Peripheral blood stem cell (PBSC) transplantation; Procedure: Allogeneic hematopoietic stem cell transplant (HSCT); Drug: Filgrastim; Genetic: T-Rapa cell Donor Lymphocyte Infusion (DLI)
- Arm IVD cohort 2 (conventional DLI) (Experimental): Patients receive low intensity fludarabine phosphate IV and cyclophosphamide IV on days -6 to -3. Patients undergo DLI with unmanipulated donor T-cells on day 14 (single T- cell DLI in patients with low CD4 count between 100 and 200 inclusive)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Peripheral blood stem cell (PBSC) transplantation; Genetic: T cell donor lymphocyte infusion (DLI) with unmanipulated donor T cells; Procedure: Allogeneic hematopoietic stem cell transplant (HSCT); Drug: Filgrastim
- Arm IVD cohort 3 (multiple Th2 DLI) (Experimental): Patients with nonlymphoma diagnosis or rapidly progressive lymphoma undergo DLI with multiple infusions of sirolimus generated donor Th2 cells beginning on day 14 (multiple T-Rapa cell DLI in patients with CD4 count lower than 100 or ALC lower than 300)
  Interventions: Drug: Rituximab; Drug: Fludarabine; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Procedure: Peripheral blood stem cell (PBSC) transplantation; Drug: Prednisone; Procedure: Allogeneic hematopoietic stem cell transplant (HSCT); Drug: Filgrastim; Genetic: T-Rapa cell Donor Lymphocyte Infusion (DLI)
- Arm IVA (12-day expanded Th2 DLI) (Experimental): Patients receive low-intensity preparative chemotherapy with fludarabine phosphate IV and cyclophosphamide IV on days -6 to -3, cyclosporine by mouth twice a day (PO BID) on days -4 to 100, and standard dose sirolimus PO on days -2 to 14. Patients undergo mobilized allogeneic peripheral blood stem cells (PBSC) on day 0. Patients undergo DLI with 12-day expanded sirolimus-generated donor Th2 cells on day 14.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Peripheral blood stem cell (PBSC) transplantation; Genetic: T cell donor lymphocyte infusion (DLI) with unmanipulated donor T cells; Procedure: Allogeneic hematopoietic stem cell transplant (HSCT); Drug: Filgrastim
- Arm IVB (6-day expanded Th2 DLI) (Experimental): Patients receive low-intensity preparative chemotherapy with fludarabine phosphate IV and cyclophosphamide IV on days -6 to -3, cyclosporine PO BID on days -4 to 100, and standard dose sirolimus PO on days -2 to 14. Patients undergo mobilized allogeneic PBSC or bone marrow transplant on day 0. Patients undergo DLI with 6-day expanded sirolimus-generated donor Th2 cells on day 14.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Peripheral blood stem cell (PBSC) transplantation; Genetic: T cell donor lymphocyte infusion (DLI) with unmanipulated donor T cells; Procedure: Allogeneic hematopoietic stem cell transplant (HSCT); Drug: Filgrastim
- Arm IVC (6-day expanded Th2 DLI and High-Dose Sirolimus) (Experimental): Patients receive low-intensity preparative chemotherapy with fludarabine phosphate IV and cyclophosphamide IV on days -6 to -3, cyclosporine PO BID on days -7 to 100 and high dose sirolimus PO on days -4 to 7, Patients undergo mobilized allogeneic PBSC on day 0. Patients undergo DLI with 6-day expanded sirolimus-generated donor Th2 cells on day 14.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Peripheral blood stem cell (PBSC) transplantation; Genetic: T cell donor lymphocyte infusion (DLI) with unmanipulated donor T cells; Procedure: Allogeneic hematopoietic stem cell transplant (HSCT); Drug: Filgrastim

INTERVENTIONS:
Drug: Rituximab — Rituximab: 375 mg/m(2)/day intravenous (IV), day 1 (for cluster of differentiation 20 (CD20+) patients).
  Other Names: Rituxan
  Arms: Arm IVD cohort 3 (multiple Th2 DLI)
Drug: Fludarabine — Fludarabine: 30 mg/m(2)/day intravenous (IV), days -6 to -3.
  Other Names: Fludara
Drug: Etoposide — Etoposide: 50 mg/m(2)/day continuous intravenous (CIV), days 1-4.
  Other Names: Toposar
  Arms: Arm IVD cohort 3 (multiple Th2 DLI)
Drug: Doxorubicin — Doxorubicin:10 mg/m(2)/day continuous intravenous (CIV), days 1-4.
  Other Names: Doxil
  Arms: Arm IVD cohort 3 (multiple Th2 DLI)
Drug: Vincristine — Vincristine: 0.4 mg/m(2)/day continuous intravenous (CIV), days 1-4.
  Other Names: Leurocristine
  Arms: Arm IVD cohort 3 (multiple Th2 DLI)
Drug: Cyclophosphamide — Cyclophosphamide, 300 mg/m(2)/day intravenous (IV), days -6 to -3.
  Other Names: Cytoxan
Procedure: Peripheral blood stem cell (PBSC) transplantation — PBSC transplantation, peripheral blood progenitor cell transplantation, transplantation, peripheral blood stem cell.
Genetic: T cell donor lymphocyte infusion (DLI) with unmanipulated donor T cells — The dose of the T cells will attempt to be held constant for each study recipient (target dose 2.5 x 10(7) T cells/kg; minimum dose will be 1 x 10(7) T cells/kg).
  Arms: Arm IVA (12-day expanded Th2 DLI); Arm IVB (6-day expanded Th2 DLI); Arm IVC (6-day expanded Th2 DLI and High-Dose Sirolimus); Arm IVD cohort 2 (conventional DLI)
Drug: Prednisone — Prednisone: 60 mg/m(2)/day by mouth (PO), days 1-5.
  Other Names: Deltasone
  Arms: Arm IVD cohort 3 (multiple Th2 DLI)
Procedure: Allogeneic hematopoietic stem cell transplant (HSCT) — Allogeneic Hematopoietic Stem Cell Transplant.
Drug: Filgrastim — Filgrastim: 5 mcg/kg/day subcutaneous (SC), day 6 (require absolute neutrophil count (ANC) > 1000, two values; or ANC > 5000 cells/ul on one occasion).
  Other Names: Neupogen
Genetic: T-Rapa cell Donor Lymphocyte Infusion (DLI) — The dose of T helper 2 (Th2) cells or unmanipulated donor T cells will attempt to be held constant for each study recipient (target dose 2.5 x 10(7) Th2/kg; minimum dose will be 1 x 10(7) Th2/kg).
  Arms: Arm IVD cohort 1 (Th2 DLI); Arm IVD cohort 3 (multiple Th2 DLI)

SUMMARY:
Background:

Patients with cancers of the blood and immune system often benefit from transplants of stem cells from a genetically well-matched sibling. However, severe problems may follow these transplants because of the high-dose chemotherapy and radiation that accompany the procedure. Also, donated immune cells sometimes attack healthy tissues in a reaction called graft-versus-host disease (GVHD), damaging organs such as the liver, intestines and skin. To reduce toxicity of high-dose preparative chemotherapy, this study performs allogeneic transplant after low doses of chemotherapy. In an attempt to improve anti-tumor effects without increasing GVHD, this study uses donor immune cells (T helper 2 (Th2) cells) grown in the laboratory; some patients will receive standard donor immune cells (not grown in laboratory). All patients will receive immune modulating drugs sirolimus and cyclosporine to prevent GVHD.

Objective:

To determine the safety, treatment effects and rate of GVHD in patients receiving transplants that use low-intensity chemotherapy, sirolimus plus cyclosporine, and transplant booster with either Th2 cells or standard immune cells.

Eligibility:

Patients 16 to 75 years of age with acute or chronic leukemia, non-Hodgkin's lymphoma, Hodgkin's disease, multiple myeloma, or myelodysplastic syndrome.

Patients must have a suitable genetically matched sibling donor and adequate kidney, heart and lung function.

Design: The protocol has three treatment groups: cohort 1, Th2 booster at two weeks post-transplant; cohort 2, standard T cell booster at two weeks post-transplant; cohort 3, multiple infusion of Th2 cells.

Condition: Hematologic Neoplasms, Myeloproliferative Disorders

Intervention: Biological; therapeutic allogeneic lymphocytes

Drug: Sirolimus

Study Type: Interventional

Study Design: Primary Purpose: Treatment

Phase: Phase II

DETAILED DESCRIPTION:
Background

In protocol 99-C-0143, we evaluated a new approach to allogeneic hematopoietic stem cell transplant (HSCT) that involved intensive host T cell ablation and graft augmentation with in vitro generated donor T helper 2 (Th2) cells. Rapid full donor engraftment occurred with this regimen; however, grade II to IV acute graft versus host disease (GVHD) was not significantly reduced in Th2 cell recipients. In an attempt to improve clinical results using Th2 cell graft engineering, this second-generation Th2 cell clinical trial was developed that incorporates the following interventions: (1) In an attempt to reduce transplant-related toxicity, this protocol now uses a very low-intensity host preparative chemotherapy; (2) In an attempt to reduce GVHD, this study will utilize Th2 cells expanded in the presence of the immune modulation agent, rapamycin (sirolimus), as murine Th2 cells grown in rapamycin reduce GVHD more effectively than control Th2 cells; (3) To further reduce GVHD, subjects will receive a short-course of sirolimus therapy in addition to standard cyclosporine GVHD prophylaxis; and (4) Using this novel low-intensity transplant platform, compare in a preliminary manner the post-transplant outcome of patients receiving pre-emptive donor lymphocyte infusion (DLI) using either Th2 cells or unmanipulated donor T cells.

Objectives

In the setting of human leukocyte antigen (HLA)-matched sibling allogeneic HSCT using GVHD prophylaxis of cyclosporine and short-course sirolimus, compare in a preliminary manner the safety, feasibility, alloengraftment, clinical anti-tumor effects, and GVHD rate of low-intensity Preparative Chemotherapy with pre-emptive DLI using either Th2 cells or unmanipulated T cells at day 14 post-HSCT.

Eligibility

Subjects that are 16 to 75 years of age that have a suitable 6/6 HLA-matched sibling donor are potentially eligible. Subjects with a diagnosis of acute or chronic leukemia, non-Hodgkin's lymphoma, Hodgkin's disease, multiple myeloma, or myelodysplastic syndrome are potentially eligible. Adequate kidney, cardiac, and pulmonary function are required.

Design

* Patients age 18 or older with lymphoma (all types) or chronic lymphocytic leukemia will be randomized just prior to the transplant regimen to receive DLI with either donor Th2 cells (cohort 1) or unmanipulated T cells (cohort 2); n=10 patients will be accrued to each arm provided that stopping rules pertaining to excessive GVHD or graft rejection are not met. For these randomized patients, the preparative regimen will consist of low-intensity fludarabine (120 mg/m(2)) plus cyclophosphamide (1200 mg/m(2)) and GVHD prophylaxis will consist of short-course, high-dose sirolimus followed by maintenance cyclosporine. Cohorts 1 and 2 will be compared in a preliminary manner with respect to their post-transplant outcome, in particular: (a) conversion of mixed chimerism to predominant donor chimerism; (b) rate and severity of classical acute and late acute GVHD at the day 100 and day 180 post-transplant time points; and (c) time to induction of leukemia/lymphoma remission (if entering transplant with disease) or time to relapse (if entering transplant in remission).
* Patients with non-lymphoma diagnoses, patients with lymphoma that are under the age of 18 and lymphoma patients that are projected to be unable to complete the protocol-defined therapy through day 180 post-transplant will not be randomized but will be treated on cohort 3 (n=40), which will evaluate transplantation without the Flu/Cy preparative regimen and with pre-emptive Th2 cell DLI. The primary objective of cohort 3 is to evaluate whether transplantation without a preparative regimen will reduce the rate of acute GVHD associated with Th2 cell DLI from 41% (the rate observed with the fludarabine/cyclophosphamide (Flu/Cy) preparative regimen) to a rate of 15% (6 cases out of 40).

ELIGIBILITY:
* INCLUSION CRITERIA: PATIENT RECIPIENT

  1. Patients with hematologic malignancies, myelodysplasia, or myeloproliferative disorders, as summarized in the following table. The diagnosis must be histologically confirmed by the Laboratory of Pathology of National Cancer Institute (NCI) or Hackensack (There will be no central pathology review).
  2. Chronic Lymphocytic Leukemia - Disease Status: a) Relapse post-fludarabine, b) Non-Complete Response (CR) after salvage regimen.

     Hodgkin's and Non-Hodgkin's Lymphoma (all types, including Mantle Cell Lymphoma) - Disease Status: a) Primary treatment failure, b) Relapse after autologous stem cell transplant (SCT), c) Non-CR after salvage regimen

     Special Cases of High-Risk Lymphoma, including but not limited to : (1) plasma dendritic cell type, 2) Hepato-splenic T cell type, 3) gamma delta pinniculitic T cell type, 4) Muco-cutaneous natural killer (NK) cell type and 5) stage III-IV nasal NK cell type- Disease Status: a) Primary treatment failure, b) Relapse after autologous, c) Non-CR after salvage regimen, d) In first CR or any later CR

     Chronic Epstein Barr Virus (EBV)-associated lymphoproliferative disease a) At any point after diagnosis, including up-front therapy

     Multiple Myeloma - Disease Status: a) Primary treatment failure, b) Relapse after autologous stem cell transplant (SCT), c) Non-CR after salvage regimen.

     Acute Myelogenous Leukemia - Disease Status: a) CR number 1 and high-risk [excludes t(8;21), t(15;17), or inv(16)], b) CR number 2 or greater).

     Acute Lymphocytic Leukemia - Disease Status: a) CR number 1 plus high-risk [t(9;22) or bcr-abl(+); t(4;11), 1(1;19), t(8;14)], b) In CR number2 or greater.

     Myelodysplastic Syndrome - Disease Status: a) Refractory Anemia with Excess Blasts (RAEB), b) Refractory Anemia with Excess Blasts in Transformation (RAEB-T) (requires marrow and blood blasts less than 10% after induction chemotherapy).

     Myeloproliferative disorders - Disease Status: a) Idiopathic myelofibrosis, b) Polycythemia vera, c) Essential thrombocytosis, d) Chronic myelomonocytic leukemia.

     Chronic Myelogenous Leukemia (CML) - Disease Status: a) Chronic phase CML, refractory to imatinib treatment b) Accelerated phase CML. b) Accelerated phase CML

     Patients with myeloproliferative disorders must be end-stage, which is primarily defined as disease severity refractory to splenectomy.
  3. Patient age of 16 to 75 years.
  4. Consenting first degree relative matched at 6/6 HLA antigens (A, B, and DR).
  5. Patient or legal guardian must be able to give informed consent.
  6. All previous intravenous therapy administered outside of the National Institutes of Health (NIH) Clinical Center must be completed at least 2 weeks prior to study entry, with recovery to less than or equal to non-hematologic grade 2 toxicity of previous therapy.
  7. Eastern Cooperative Oncology Group (ECOG) performance status equal to 0 or 1.
  8. Life expectancy of at least 3 months.
  9. Patients with acute leukemia must have chemotherapy sensitive disease, as defined by at least a 50% reduction in circulating absolute blast count due to the most proximal regimen.
  10. Left ventricular ejection fraction greater than or equal to 45%, preferably by 2-dimension (2-D) echo, or by multi-gated acquisition scan (MUGA). However, patients with left ventricular ejection fraction (LVEF) of between 35% and 44% may also be eligible provided that such patients are cleared by a Cardiology Consultation that must include a cardiac stress test.
  11. Corrected diffusing capacity or transfer of the lung for carbon monoxide (DLCO) greater than 50% of expected value.
  12. Creatinine less than or equal to 1.5 mg/dl or creatinine clearance greater than or equal to 50 ml/min.
  13. Serum total bilirubin less than 2.5 mg/dl; serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) equal 2.5 times upper limit of normal. Values above these levels may be accepted, at the discretion of the principal investigator (PI) or study chairman, if such elevations are thought to be due to liver involvement by malignancy or graft versus host disease (GVHD).
  14. Adequate central venous access potential.
  15. Potential patients referred for the study may not be eligible for the experimental protocol therapy due to reasons such as uncertainty about donor human leukocyte antigen (HLA) typing or need to control malignant disease, infection, or metabolic abnormality such as hypercalcemia on a emergent basis. Should a referred patient present to us in such a scenario, the patient will be referred back to their primary hematologist-oncologist for treatment. However, if referral back to the referring physician is not in the best interest of the patient according to the clinical judgement of the principal investigator (PI), then the patient may receive standard treatment for the malignant disease or complicating conditions (infection, metabolic problems under the current study. In other cases, a patient may have reasonable control of malignancy but does not meet the cluster of differentiation 4 (CD4) cell cut-off of 50 cells per microliter required for cohort 3 therapy; in such cases, standard care chemotherapy regimens may be administered for the specific goal of reducing the CD4 count (that is, immune depleting regimens such as the pentostatin plus cyclophosphamide combination, administered similar to the manner that we have developed on protocol 08-C- 0088). If it becomes apparent that the patient will not be able to proceed to experimental therapy, then he/she must come off study. Recipient-Subjects receiving a standard therapy, and availability of receiving the same treatment elsewhere, outside of a research protocol. Because such standard care therapy is not experimental, it is not necessary to complete the eligibility criteria prior to receiving such standard care; however, prior to initiation of the experimental therapy, the patient must meet each of the eligibility criteria detailed above. Attempts will be made to standardize such pretransplant chemotherapy (by administration of etoposide, prednisolone, oncovin, cyclophosphamide, hydroxydaunorubicin, fludarabine, rituximab (EPOCH-FR) chemotherapy, which is detailed later in this protocol); however, other regimens using approved agents will be allowed if such regimens are thought to be in the best interest of the patient.

INCLUSION CRITERIA: DONOR

1. First-degree relative with genotypic identity at 6/6 HLA loci (HLA- A, B, and DR).
2. Age 11 to 90 years and able to give consent or assent. For donors < 18 years old, the legal guardian must be able to provide informed consent.
3. Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.
4. Donors must be human immunodeficiency virus (HIV) negative.
5. Donors with a history of hepatitis B or hepatitis C infection may be eligible. However, eligibility determination of such patients will require a hepatology consultation. The risk/benefit of the transplant and the possibility of transmitting hepatitis will be discussed with the patient and eligibility will then be determined by the principal investigator and lead associate investigator (LAI).
6. Lactating donors must substitute formula feeding for her infant during period of filgrastim administration (to prevent any filgrastim effect on infant).

EXCLUSION CRITERIA: PATIENT

1. Active infection that is not responding to antimicrobial therapy.
2. Active central nervous system (CNS) involvement by malignancy.
3. HIV infection (treatment may result in progression of HIV and other viral infections).
4. Chronic active hepatitis B. Patient may be hepatitis B core antibody positive. For patients with concomitant positive hepatitis B surface antigen, patient will require a hepatology consultation. The risk/benefit profile of transplant and hepatitis B will be discussed with the patient and eligibility determined by the principal investigator and Lead Associate Investigator.
5. Hepatitis C infection. Patient may have hepatitis C infection. However, each patient will require a hepatology consultation. The risk/benefit profile of transplant and hepatitis C will be discussed with the patient and eligibility determined by the principal investigator and Lead Associate Investigator.
6. Pregnant or lactating. Patients of childbearing potential must use an effective method of contraception. The effects of the chemotherapy, the subsequent transplant and the medications used after the transplant are highly likely to be harmful to a fetus. The effects upon breast milk are also unknown and may be harmful to the infant.
7. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.

EXCLUSION CRITERIA: DONOR

1. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.
2. History of hypertension that is not controlled by medication, stroke, autoimmune disease, or severe heart disease (donors with symptomatic angina will be excluded). Donors with a history of coronary artery bypass grafting or angioplasty who are symptom free will receive a cardiology evaluation and be considered on a case-by-case basis.
3. History of prior malignancy. However, cancer survivors who have undergone potentially curative therapy may be considered for stem cell donation on a case-by-case basis. In addition, donors with localized cancer such as prostate cancer that are on a watch-and-wait management due to the low-risk of disease progression may also be considered for stem cell donation on a case-by-case basis. The risk/benefit of the transplant and the possibility of transmitting viable tumor cells at the time of transplantation will be discussed with the patient.
4. Donors must not be pregnant (unknown effect of filgrastim on fetus). Donors of childbearing potential must use an effective method of contraception.
5. Anemia (Hemoglobin (Hb) less than 11 gm/dl) or thrombocytopenia (platelets less than 100,000 per microliter). However, potential donors with Hb levels less than 11 gm/dl that is due to iron deficiency will be eligible as long as the donor is initiated on iron replacement therapy and the case is individually approved by National Institutes of Health (NIH) or Hackensack Blood Bank.

Ages: 11 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage JO. Bone marrow transplantation. N Engl J Med. 1994 Mar 24;330(12):827-38. doi: 10.1056/NEJM199403243301206. No abstract available. PMID 8114836
- [Background] Jamshed S, Fowler DH, Neelapu SS, Dean RM, Steinberg SM, Odom J, Bryant K, Hakim F, Bishop MR. EPOCH-F: a novel salvage regimen for multiple myeloma before reduced-intensity allogeneic hematopoietic SCT. Bone Marrow Transplant. 2011 May;46(5):676-81. doi: 10.1038/bmt.2010.173. Epub 2010 Jul 26. PMID 20661232
- [Result] Fowler DH, Mossoba ME, Steinberg SM, Halverson DC, Stroncek D, Khuu HM, Hakim FT, Castiello L, Sabatino M, Leitman SF, Mariotti J, Gea-Banacloche JC, Sportes C, Hardy NM, Hickstein DD, Pavletic SZ, Rowley S, Goy A, Donato M, Korngold R, Pecora A, Levine BL, June CH, Gress RE, Bishop MR. Phase 2 clinical trial of rapamycin-resistant donor CD4+ Th2/Th1 (T-Rapa) cells after low-intensity allogeneic hematopoietic cell transplantation. Blood. 2013 Apr 11;121(15):2864-74. doi: 10.1182/blood-2012-08-446872. Epub 2013 Feb 20. PMID 23426943
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0055.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was 442 (221 donors; 221 patients). 57 recipients were treated on cohorts no longer in the protocol due to amendments. Thus, 164 of 221 recipient data is presented. No patients were eligible for therapy on arm IVD, cohort 2.
Groups:
- Arm IVD Cohort 1 (Th2 DLI): Patients receive low intensity fludarabine phosphate intravenous (IV) and cyclophosphamide IV on days -6 to -3. Patients undergo donor lymphocyte infusion (DLI) with sirolimus generated donor T-helper 2 (Th2) cells on day 14 (single T-Rapa cell DLI in patients with cluster of differentiation 4 (CD4) count between 100 and 200 inclusive).
  Etoposide: Etoposide: 50 mg/m(2)/day continuous intravenous (CIV), days 1-4
  Doxorubicin: Doxorubicin:10 mg/m(2)/day CIV, days 1-4
  Vincristine: Vincristine:0.4 mg/m(2)/day CIV, days 1-4
  Cyclophosphamide: Cyclophosphamide, 750 mg/m(2)/day IV, day 5
  T cell donor lymphocyte infusion (DLI) with sirolimus generated donor TH-2 cells: The cell of the Th2 cells will attempt to be held constant for each study receipient (target dose 2.5 x 107 Th2/kg; minimum dose will be 1 x 107 Th2/kg).
- Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus): Patients receive low-intensity preparative chemotherapy with fludarabine phosphate IV and cyclophosphamide IV on days -6 to -3, cyclosporine PO BID on days -7 to 100 and high dose sirolimus PO on days -4 to 7, Patients undergo mobilized allogeneic PBSC on day 0. Patients undergo DLI with 6-day expanded sirolimus-generated donor Th2 cells on day 14.
- Healthy Donors: Donate donor immune cells for recipients.
  No data was collected from the donor population.
Period: Overall Study
Arm/Group | Arm IVD Cohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus) | Healthy Donors
Started | 1 | 34 | 40 | 44 | 45 | 221
Completed | 1 | 27 | 40 | 44 | 42 | 221
Not Completed | 0 | 7 | 0 | 0 | 3 | 0
Not completed — Progressive malignancy | 0 | 7 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment was 442 (221 donors; 221 patients). No data was collected from the donor population. 57 recipients were treated on cohorts no longer in the protocol due to amendments. Thus, 164 of 221 recipient data is presented. No patients were eligible for therapy on arm IVD, cohort 2.
Groups:
- Arm IVDcohort 1 (Th2 DLI): Patients receive low intensity fludarabine phosphate intravenous (IV) and cyclophosphamide IV on days -6 to -3. Patients undergo donor lymphocyte infusion (DLI) with sirolimus generated donor T-helper 2 (Th2) cells on day 14 (single T-Rapa cell DLI in patients with cluster of differentiation 4 (CD4) count between 100 and 200 inclusive).
- Total: Total of all reporting groups
Arm/Group | Arm IVDcohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus) | Total
Number analyzed (Participants) | 1 | 34 | 40 | 44 | 45 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 33 | 36 | 41 | 42 | 153
  >=65 years | 0 | 1 | 4 | 3 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 | 45.96 (12.41) | 49.68 (12.92) | 47.66 (12.45) | 50.19 (13.50) | 49.44 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 17 | 21 | 13 | 59
  Male | 1 | 26 | 23 | 23 | 32 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 11 | 8 | 10 | 4 | 33
  Not Hispanic or Latino | 1 | 23 | 32 | 34 | 41 | 131
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 4 | 2 | 4 | 11
  White | 1 | 20 | 28 | 30 | 36 | 115
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 11 | 8 | 10 | 4 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 34 | 40 | 44 | 45 | 164

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients to Receive T Cell Infusion
Description: T cells administered by intravenous infusion after patient received transplant.
Time Frame: first 100 days post-transplant
Measure: Number; unit: percentage of patients
Arm/Group | Arm IVD Cohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus)
Number analyzed (Participants) | 1 | 27 | 40 | 44 | 42
percentage of patients | 100 | 100 | 100 | 100 | 100

2. Primary Outcome: Percentage of Patients With ≥ Grade 2 Acute Graft Versus Host Disease (GVHD)
Description: GVHD of the skin, liver and gut were graded on a scale of 1, 2, 3, and 4 (e.g. the grades are not added together) using the National Institutes of Health Consensus Criteria. Grade 1 is minimal GVHD, Grade 2 is moderate GVHD, Grade 3 is severe GVHD and Grade 4 is very severe GVHD. Grade 4 is a worse outcome than Grade 1.
Time Frame: first 100 days post-transplant
Measure: Number; unit: percentage of patients
Arm/Group | Arm IVD Cohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus)
Number analyzed (Participants) | 1 | 27 | 40 | 44 | 42
percentage of patients | 0 | 11.11 | 10 | 40.91 | 40.48

3. Secondary Outcome: Detection of of Post-transplantation Cluster of Differentiation 4 (CD4)+ and CD8+ T-cell Production of T Helper 1 -2 (Th1-Th2)-Type Cytokines
Description: Detection of cytokine secretion was done by enzyme-linked immunosorbent assay.
Time Frame: First 100 days post-transplant
Population: This outcome measure was not done. Data was not collected for this outcome measure due to premature closure of study.
Arm/Group | Arm IVD Cohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Patients With Opportunistic Infection
Description: Participants are susceptible to opportunistic infections such as bacterial, fungal, viral, protozoan infections and more due to immune suppression from chemotherapy drugs used to treat their disease.
Time Frame: First 100 days post-transplant
Measure: Number; unit: percentage of participants
Groups:
- Arm IVB (6-day Expanded Th2 DLI): Arm IVB Patients receive low-intensity preparative chemotherapy with fludarabine phosphate IV and cyclophosphamide IV on days -6 to -3, cyclosporine PO BID on days -4 to 100, and standard dose sirolimus PO on days -2 to 14. Patients undergo mobilized allogeneic PBSC or bone marrow transplant on day 0. Patients undergo DLI with 6-day expanded sirolimus-generated donor Th2 cells on day 14.
Arm/Group | Arm IVD Cohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus)
Number analyzed (Participants) | 1 | 27 | 40 | 44 | 42
percentage of participants | 0 | 11.11 | 7.50 | 9.09 | 11.90

5. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm IVD Cohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus)
Number analyzed (Participants) | 1 | 27 | 40 | 44 | 42
Participants | 1 | 27 | 40 | 44 | 42

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 5 years.
Description: Enrollment was 442 (221 donors; 221 patients). No data was collected from the donor population. 57 recipients were treated on cohorts no longer in the protocol due to amendments. Thus, 164 of 221 recipient data is presented. No patients were eligible for therapy on arm IVD, cohort 2.
Arm/Group | Arm IVD Cohort 1 (Th2 DLI) | Arm IVD Cohort 3 (Multiple Th2 DLI) | Arm IVA (12-day Expanded Th2 DLI) | Arm IVB (6-day Expanded Th2 DLI) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus)
All-Cause Mortality (participants affected / at risk) | 0/1 | 14/34 | 22/40 | 24/44 | 22/45
Serious Adverse Events (participants affected / at risk) | 1/1 | 22/34 | 37/40 | 35/44 | 31/45
Other Adverse Events (participants affected / at risk) | 1/1 | 28/34 | 40/40 | 38/44 | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm IVD Cohort 1 (Th2 DLI) (N=1) | Arm IVD Cohort 3 (Multiple Th2 DLI) (N=34) | Arm IVA (12-day Expanded Th2 DLI) (N=40) | Arm IVB (6-day Expanded Th2 DLI) (N=44) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus) (N=45)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 5 (10) | 4 (6) | 16 (25) | 5 (18)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 1 (1) | 4 (10) | 12 (16) | 1 (2)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bilirubin (hyperbilirubinemia) (Nervous system disorders) | 0 (0) | 3 (4) | 6 (7) | 7 (8) | 0 (0)
Blood/Bone Marrow - Other (engraftment syndrome) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrhythmia - Other (atrial fibrillation) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac General - Other (congestive heart failure) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I (cTnI) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 7 (7) | 7 (7)
Conduction abnormality/atrioventricular heart block::AV Block-First degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conduction abnormality/atrioventricular heart block::AV Block-Second degree Mobitz Type II (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 0 (0) | 0 (0) | 3 (8) | 4 (4) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Death not associated with CTCAE term::Death NOS (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 5 (5)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 0 (0) | 7 (8) | 9 (9) | 12 (12) | 11 (11)
Death not associated with CTCAE term::Multi-organ failure (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term::Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (skin thickening of chest, abdomen, back of legs and shoulders for the past 3-4 mon)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 10 (10) | 16 (16) | 11 (11)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 1 (1)
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema: head and neck (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 10 (11) | 25 (25) | 5 (5) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 1 (1) | 14 (14) | 10 (10) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal - Other (Abdominal pain (GVHD of the gut) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (abdominal pain, nausea and diarrhea c/w GVHD) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 8 (14) | 10 (16) | 3 (4)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI::Lower GI NOS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hemorrhage, GI::Upper GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage/Bleeding - Other (Conjunctival, low platelet ct) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (Massive Intracranial hemorrhage of left frontal lobe mass) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage/Bleeding - Other (diffuse alveolar hemorrhage) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 6 (7) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 12 (13) | 11 (11) | 3 (3)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Abdomen NOS
Infection (documented clinically (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Bladder (urinary)
Infection (Infections and infestations) | 0 (0) | 8 (9) | 5 (6) | 13 (13) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Bronchus
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) — (ANC <1.0 x 10e9/L)::Catheter-related
Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Colon
Infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 12 (12) | 2 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Meninges (meningitis)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Mucosa
Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Nose
Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Rectum
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Sinus
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Skin (cellulites)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Stomach
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Ungual (nails)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Upper aerodigestive NOS
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Upper airway NOS
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection - Other (C.Diff: PCR +) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - Other (HHV6 reactivation; admitted for anemia & leukocytosis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Influenza A +) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - Other (R. wrist septic arthritis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (pseudomonas bacteremia/sepsis.) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (worsening right great toe pain with drainage and now neutropenic) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Appendix (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1) | 13 (14) | 10 (11) | 18 (22) | 13 (13)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bone (osteomyelitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Brain (encephalitis, infectious) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Brain + Spinal cord (encephalomyelitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 4 (4) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 1 (1) | 1 (1) | 7 (7) | 8 (8) | 6 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils::External ear (otitis externa) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 0 (0) | 4 (4) | 12 (13) | 24 (24) | 11 (11)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lymphatic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Peritoneal cavity (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pleura (empyema) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Rectum (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils::Stomach (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 4 (4) | 6 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with unknown ANC::Abdomen NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Infection with unknown ANC::Meninges (meningitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC::Sinus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection with unknown ANC::Upper aerodigestive NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Leukocytes (total WBC) (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic/Laboratory - Other (ph>7.5 with life threating consequences ALKALOSIS) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic/Laboratory - Other (steroid induced hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4) | 5 (5) | 1 (1)
Neuropathy: cranial::CN III Pupil, upper eyelid, extra ocular movements (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neuropathy: cranial::CN VI Lateral deviation of eye (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 3 (3) | 15 (21) | 13 (20) | 7 (10)
Obstruction, GI::Gallbladder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstruction, GI::Small bowel NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstruction/stenosis of airway::Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction/stenosis of airway::Trachea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular/Visual - Other (GVHD) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular/Visual - Other (ocular GVHD, restasis started; EXTENSIVE CGVHD) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Pain::Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Perforation, GI::Small bowel NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 1 (1)
Platelets (Investigations) | 0 (0) | 2 (3) | 7 (8) | 7 (18) | 3 (9)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (6) | 5 (5) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 5 (6) | 0 (0)
Prolonged QTc interval (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 11 (11) | 9 (9) | 4 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 2 (2)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secondary Malignancy - (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — possibly related to cancer treatment (basal cell carcinoma (left supraclavicular). Start/end date is approx.)
Secondary Malignancy - possibly related to cancer treatment (squamous cell carcinoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (squamous cell carcinoma of skin x2 (forehead and left arm). Resolve date approx.)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (3) | 3 (3) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stricture/stenosis (including anastomotic), GU::Urethra (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia::Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ulcer, GI::Stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm IVD Cohort 1 (Th2 DLI) (N=1) | Arm IVD Cohort 3 (Multiple Th2 DLI) (N=34) | Arm IVA (12-day Expanded Th2 DLI) (N=40) | Arm IVB (6-day Expanded Th2 DLI) (N=44) | Arm IVC (6-day Expanded Th2 DLI and High Dose Sirolimus) (N=45)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1) | 17 (38) | 34 (53) | 29 (81) | 36 (78)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 12 (17) | 24 (43) | 20 (27) | 24 (57)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 6 (10) | 10 (26) | 5 (7) | 9 (13)
Alkaline phosphatase (Investigations) | 0 (0) | 4 (5) | 2 (2) | 3 (3) | 1 (1)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Ascites (non-malignant) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Nervous system disorders) | 0 (0) | 8 (15) | 7 (13) | 15 (24) | 14 (35)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiac troponin I (cTnI) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Creatinine (Investigations) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Cytokine release syndrome/acute infusion reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (8) | 9 (9) | 6 (6) | 13 (13)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Dry eye syndrome (Eye disorders) | 0 (0) | 4 (4) | 7 (7) | 4 (4) | 5 (5)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Eyelid dysfunction (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (9) | 1 (1) | 3 (3) | 4 (4) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 2 (2) | 9 (12) | 10 (10) | 1 (1)
Fibrinogen (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 14 (24) | 34 (112) | 27 (53) | 18 (36)
Hemorrhage, GI::Colon (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GI::Lower GI NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GU::Bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperpigmentation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Induration/fibrosis (skin and subcutaneous tissue) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Abdomen NOS
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Anal/perianal
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Bladder (urinary)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Catheter-related
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1) — (ANC <1.0 x 10e9/L)::Colon
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Esophagus
Infection (documented clinically or microbiologically) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Gallbladder (cholecystitis)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Joint
Infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Mucosa
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Oral cavity-gums (gingivitis)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Pharynx
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Skin (cellulites)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Soft tissue NOS
Infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 4 (4) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Upper airway NOS
Infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection - Other (Specify, __) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (CMV reactivation) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Possible bronchiolitis obliterans) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Right arm pain and swelling-catheter celulitis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Sinusitis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infection - Other (Stool cultures 5/31: Yersinia, Novovirus as well as H. nana. (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 0 (0) | 15 (19) | 7 (7) | 10 (11) | 14 (14)
Infection with normal ANC or Grade 1 or 2 neutrophils::Brain (encephalitis, infectious) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils::Conjunctiva (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Dental-tooth (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 0 (0) | 5 (6) | 4 (4) | 7 (7) | 10 (10)
Infection with normal ANC or Grade 1 or 2 neutrophils::Middle ear (otitis media) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Mucosa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nerve-peripheral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nose (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Paranasal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pelvis NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Penis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Peritoneal cavity (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Rectum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Salivary gland (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 5 (6) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Stomach (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 0 (0) | 12 (14) | 9 (11) | 17 (17) | 26 (26)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 0 (0) | 9 (9) | 11 (11) | 5 (5) | 10 (10)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vagina (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Infection with unknown ANC::Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Infection with unknown ANC::Mucosa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC::Sinus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection with unknown ANC::Skin (cellulitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC::Vagina (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukocytes (total WBC) (Investigations) | 0 (0) | 0 (0) | 6 (12) | 0 (0) | 0 (0)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphedema-related fibrosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (25) | 0 (0) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 9 (15) | 16 (23) | 6 (7)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 1 (1)
Mental status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood alteration::Agitation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood alteration::Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam)::Large bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 12 (12) | 4 (4) | 3 (3)
Mucositis/stomatitis (functional/symptomatic)::Large bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-upper (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 7 (8) | 40 (136) | 37 (64) | 26 (44)
Ocular surface disease (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ocular/Visual - Other (GVHD Gd 1) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular/Visual - Other (Occular GVHD) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Worsening Rt eye swelling on 6/1: MRI orbits 6/1 showed enlargement of eyelid nodule
Ocular/Visual - Other (red and itchy eyes) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 5 (8) | 10 (12) | 9 (10) | 9 (10)
Pain - Other (jaw/scalp) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain::Abdomen NOS (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Pain::Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain::Esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pain::Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Oral-gums (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 5 (6) | 17 (39) | 16 (30) | 19 (34)
Platelets (Investigations) | 0 (0) | 7 (10) | 28 (77) | 18 (33) | 23 (41)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 5 (8) | 5 (7) | 3 (3) | 5 (7)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 7 (7) | 16 (32) | 10 (19) | 14 (21)
Prolonged QTc interval (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 2 (2)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 30 (30) | 17 (17) | 18 (18)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 2 (2)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rigors/chills (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum-high (hypernatremia) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 11 (17) | 4 (5) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste alteration (dysgeusia) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thyroid function, low (hypothyroidism) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 4 (8) | 0 (0) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
118 subjects were enrolled on this study on cohorts no longer represented in the protocol due to amendments. Of the 118, 50% were participants and 50% were donors. These participants are not represented in the data being reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT00074490/Prot_SAP_000.pdf